CLINICAL TRIAL: NCT02050828
Title: A Phase 2, Randomized, Active-Controlled, Double-Masked, Multi-Center Study to Assess the Safety and Efficacy of Daily Subcutaneous AKB-9778 Administered for 3 Months, as Monotherapy or Adjunctive to Ranibizumab, in Subjects With Diabetic Macular Edema
Brief Title: The TIME-2 Study: A Phase 2 Study of AKB-9778, a Novel Tie-2 Activator, in Patients With Diabetic Macular Edema
Acronym: TIME-2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aerpio Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AKB-9778-CI-2003
Record Dates: First submitted 2014-01-29; First posted 2014-01-31 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Diabetic Macular Edema (DME)
MeSH Terms: interventions — AKB-9778; Ranibizumab; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AKB-9778 15 mg BID monotherapy (Experimental): Subcutaneous AKB-9778 15 mg BID (total daily dose of 30 mg/day) plus monthly sham intravitreal injection for 3 months.
  Interventions: Drug: AKB-9778; Drug: Sham
- AKB-9778 15 mg BID + ranibizumab 0.3 mg (Experimental): Subcutaneous AKB-9778 15 mg BID (total daily dose of 30 mg/day) plus ranibizumab 0.3 mg monthly intravitreal injection for 3 months.
  Interventions: Drug: AKB-9778; Drug: ranibizumab
- ranibizumab 0.3 mg monotherapy (Active Comparator): Placebo subcutaneous injection (BID) plus ranibizumab 0.3 mg monthly intravitreal injection for 3 months.
  Interventions: Drug: ranibizumab; Drug: Placebo

INTERVENTIONS:
Drug: AKB-9778
  Arms: AKB-9778 15 mg BID + ranibizumab 0.3 mg; AKB-9778 15 mg BID monotherapy
Drug: ranibizumab
  Other Names: Lucentis
  Arms: AKB-9778 15 mg BID + ranibizumab 0.3 mg; ranibizumab 0.3 mg monotherapy
Drug: Placebo
  Arms: ranibizumab 0.3 mg monotherapy
Drug: Sham
  Arms: AKB-9778 15 mg BID monotherapy

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of AKB-9778 administered as daily subcutaneous injections with and without monthly intravitreal injections of ranibizumab for 3 months in patients with diabetic macular edema.

ELIGIBILITY:
The following is an abbreviated list of inclusion criteria:

* Adults between 18 to 80 years of age, inclusive
* Diagnosis of diabetes mellitus (type 1 or type 2)
* Decrease in vision in the study eye determined to be primarily the result of DME
* Definite retinal thickening due to diffuse DME involving the central macula in the study eye
* Central subfield thickness of at least 325 µm by sdOCT with presence of intraretinal fluid in the study eye
* ETDRS BCVA letter score ≤ 76 and ≥ 24 in the study eye

The following is an abbreviated list of exclusion criteria:

* Hemoglobin A1C (HbA1C) ≥ 12.0% at Screening
* History of non infectious uveitis
* Decrease in visual acuity due to causes other than DME in the study eye
* History of any of the following in the study eye (however, the following are not exclusionary in the fellow eye):

  1. Prior pars plana vitrectomy
  2. Any ocular surgery within 3 months prior to Day 1
  3. YAG capsulotomy within 3 months prior to Day 1
  4. Panretinal scatter photocoagulation (PRP) or focal laser within 3 months prior to Day 1 or anticipated need for PRP during the course of the study
  5. Prior intravitreal, subtenon, or periocular steroid therapy within 3 months prior to Day 1
  6. Prior treatment with intravitreal anti-vascular endothelial growth factor (VEGF) treatment within 8 weeks prior to Day 1

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-01; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in spectral domain optical coherence tomography (sdOCT)-measured central subfield thickness (CST) | Month 3

SECONDARY OUTCOMES:
Mean change from baseline in Early Treatment Diabetic Retinopathy Study (ETDRS) Best Corrected Visual Acuity (BCVA) | Month 3

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - Pheonix, Arizona
  - Tucson, Arizona
  - Arcadia, California
  - Bakersfield, California
  - Beverly Hills, California
  - Palm Desert, California
  - Sacramento, California
  - Santa Ana, California
  - Santa Barbara, California
  - Golden, Colorado
  - Boynton Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Miami, Florida
  - Sarasota, Florida
  - Stuart, Florida
  - Winter Haven, Florida
  - Baltimore, Maryland
  - Jackson, Michigan
  - Omaha, Nebraska
  - Reno, Nevada
  - Rochester, New York
  - Charlotte, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Portland, Oregon
  - Florence, South Carolina
  - Rapid City, South Dakota
  - Nashville, Tennessee
  - Abilene, Texas
  - Austin, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - McAllen, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Warrenton, Virginia
  - Bellevue, Washington